CLINICAL TRIAL: NCT06721832
Title: The Effect of High-thoracic Erector Spinae Plane Block on Postoperative Pain and Diaphragmatic Function in Posterior Cervical Spine Surgery: a Randomized Controlled Trial
Brief Title: The Effect of High-thoracic Erector Spinae Plane Block on Postoperative Pain and Diaphragmatic Function in Posterior Cervical Spine Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, LECTURER, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC 13-10-2024
Record Dates: First submitted 2024-11-28; First posted 2024-12-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Cervical Spine Surgery; Pain Management
Keywords: ESP; PAIN; Posterior cervical surgery
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group E (Active Comparator): patients will receive bilateral in-plane ultrasound guided erector spinea plane block with 30 ml of bupivacaine 0. 25% (15 ml in each side) after induction of general anesthesia
  Interventions: Procedure: Erector spina plane block (ESP); Drug: Bupivacain (preoperative)
- Group C (Placebo Comparator): patients will receive a sham block with saline at the corresponding puncture site and same volumes as in group E (sham block) after induction of general anesthesia
  Interventions: Procedure: Erector spina plane block (ESP)

INTERVENTIONS:
Procedure: Erector spina plane block (ESP) — The block will be performed in prone position under complete aseptic condition. The site to be blocked will be painted with 5% povidone iodine followed by 70% ethyl alcohol and draped. Linear high-frequency ultrasound probe (7 -15 mhz) (General Electric; GE, "LOGIQ E") T1 transverse process will be approached with an 18 G Tuohy's needle in caudal-to-cranial direction. A total of 30 ml of 0.25% bupivacaine was administered deep to erector spinae muscle (ESM) bilaterally.
Drug: Bupivacain (preoperative) — The block will be performed in prone position under complete aseptic condition. The site to be blocked will be painted with 5% povidone iodine followed by 70% ethyl alcohol and draped. Linear high-frequency ultrasound probe (7 -15 mhz) (General Electric; GE, "LOGIQ E") T1 transverse process will be approached with an 18 G Tuohy's needle in caudal-to-cranial direction. A total of 30 ml of 0.25% bupivacaine was administered deep to erector spinae muscle (ESM) bilaterally.
  Arms: Group E

SUMMARY:
Posterior cervical spine surgery, often performed on older individuals with significant comorbidities, is one of the most painful surgical operations. Anesthesiologists face a unique challenge in managing pain following these surgeries,Erector spinae plane block (ESPB) is a relatively novel block and was first described for chronic thoracic neuropathic pain in 2016.Cervical erector spinae plane (ESP) block has been described to anesthetize the brachial plexus (BP), however, the mechanism of its clinical effect remains unknown. As the prevertebral fascia encloses the phrenic nerves, BP and erector spinae muscles to form a prevertebral compartment, a local anesthetic injected in the cervical ESP could potentially spread throughout the prevertebral compartment

ELIGIBILITY:
Inclusion Criteria:

* (ASA )classes I and II
* patients of either sex
* above the age of 18 who will undergo posterior cervical surgery

Exclusion Criteria:

* patient's refusal to participate
* any contraindications to peripheral nerve blocks
* history of ischemic heart disease
* patients on opioids for chronic pain
* patients with significant cognitive impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | VAS scores at rest and on passive neck movement postoperatively at 0, 2, 4, 6, 8, 12, 24 and 48 hours
  Visual analogue pain score which scales from zero (no pain) to ten (unbearable pain).

SECONDARY OUTCOMES:
Postoperative Pain Over Time (Visual analogue scale ) | Baseline (preoperative), 30 minutes, 2, 6, 12, and 48 hours postoperatively
  VAS pain scores at rest will be recorded at predefined postoperative intervals to evaluate pain trajectory.
Diaphragmatic Excursion | Baseline (pre-induction), 30 minutes after recovery in PACU, and 24 hours postoperatively.
  Diaphragmatic excursion will be measured using B-mode and M-mode ultrasonography during quiet breathing. Excursion is defined as the craniocaudal displacement of the diaphragm dome during tidal respiration.
Opioid Consumption | Intraoperative period and first 24 hours postoperatively.
  Total intraoperative fentanyl consumption and cumulative morphine consumption during the first 24 postoperative hours. Time to first rescue analgesic request will also be recorded.
Pulmonary Function | Baseline (preoperative), 2 hours, and 24 hours postoperatively.
  Pulmonary function will be assessed using spirometry to record forced vital capacity (FVC) and forced expiratory volume in one second (FEV₁).
Patient Satisfaction | 48 hours postoperatively.
  Patient satisfaction with postoperative analgesia will be evaluated using a 5-point Likert scale (1 = very unsatisfied, 5 = very satisfied).
Block-Related Adverse Events | 48 hours post-operatively
  Incidence of block-related adverse events, including desaturation, dyspnea, local anesthetic systemic toxicity, hematoma, or nerve injury.
Length of Hospital Stay | 48 hours postoperatively
  Duration of postoperative hospitalization measured in days.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, ELkalyobia, Egypt

IPD SHARING:
Plan to Share IPD: No